CLINICAL TRIAL: NCT06168487
Title: Phase I Non-Randomized, Unblinded, Single-Center Trial of Oral Telmisartan Alone or Combined With Selected Standard of Care Therapies for Prostate Cancer
Brief Title: Telmisartan in Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tyler J Curiel (Other)
Responsible Party: Sponsor-Investigator, Tyler J Curiel, Professor of Medicine, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY02002057; NCI-2024-07041 (Other: NCI)
Record Dates: First submitted 2023-12-04; First posted 2023-12-13 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1: Telmisartan Alone (Experimental): Patients will receive telmisartan alone.
  Interventions: Drug: Telmisartan
- Cohort 2: Telmisartan + Standard of Care Regimen (Experimental): Patients will receive telmisartan with cabazitaxel or docetaxel without abiraterone), or telmisartan with docetaxal with abirateron or olaparib or rucaparib, or talazoparib plus enzalutamide.
  Interventions: Drug: Telmisartan; Other: Standard of Care Regimen

INTERVENTIONS:
Drug: Telmisartan — Patients will be given telmisartan alone or with standard of care chemotherapy.
  Other Names: Micardis
Other: Standard of Care Regimen — Standard of Care Regimen
  Arms: Cohort 2: Telmisartan + Standard of Care Regimen

SUMMARY:
The goal of this clinical trial is to learn about the tolerability of telmisartan in patients with prostate cancer, but evidence for treatment efficacy will also be gathered.

DETAILED DESCRIPTION:
The primary objective of this study is to test the tolerability of oral telmisartan given as a single agent or combined with specific standard of care agents in selected participants with PC. Patients will be defined as tolerating telmisartan if they maintain systolic blood pressure >110 mm Hg and are without greater than grade 2 toxicities as defined in the Common Terminology Criteria for Adverse Events v5.1 for at least 60 days total telmisartan treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥18 years of age.
* Participants must be able and willing to provide informed consent or have a surrogate capable of providing same.
* Participants must not require immediate change in SOC treatment, i.e., patients with stable PSA (do not meet PCWG310 criteria for PSA progression), or with rising PSA but they remain on SOC treatment (defined as having met PCWG3 criteria for PSA progression, but do not have clinical/radiographic progression and have not met criteria for an immediate change in therapy based on PSA doubling time) as determined by their primary oncologist
* Participants must be receiving or likely to receive one of the following SOC agents for PC:

cabazitaxel, docetaxel (alone or plus abiraterone) olaparib, rucaparib, or talazoparib plus enzalutamide

* Participants must have
* ECOG performance status of 0-2
* Adequate hepatic (SCOT ≤3x ULN) and renal function (serum creatinine ≤2.5 or estimated GFR >30 cc/min)
* Standing systolic blood pressure >/= 110mm Hg
* If not on active surveillance, patient mut have castrate level testosterone
* No contraindication to telmisartan, including ACE inhibitor use in the 6 weeks prior to projected telmisartan start on trial
* All participants must have a systolic blood pressure >110 mm Hg during study enrollment assessment and throughout the study
* If participants are concurrently treated for hypertension, they must be able to allow telmisartan in addition to, or replacing their antihypertensive regimen
* Participants must be able to withstand planned research phlebotomies (Hb >10 gm/dl).
* Participants must have a blood prostate specific antigen > 1 ng/ml at study entry using the Roche Cobas immunoassay.
* Participants must be able to take or have taken their own blood pressure per the study protocol (daily during telmisartan escalation and for two weeks after the final escalation and weekly thereafter for the following month and then monthly) if normotensive at enrollment.

Exclusion Criteria:

Participants who fall into one of the following categories will NOT be eligible for this study:

* Angiotensin l receptor blocker use currently or within the 30 days prior to day 1, cycle 1.
* Patients with hypertensive urgency or emergency as defined in N Engl J Med. 2019 Nov 7;381(19):1843-1852. doi:10.1056/NEJMep1901117
* Patients who are incarcerated or homeless
* Patients who are receiving PC-specific treatment aside from cabazitaxel, docetaxel, olaparib, rucaparib, abiraterone or talazoparib plus enzalutamide or have plans to undergo the same during the study period, except local irradiation therapy to PC lesions.
* Patients on lithium therapy in any form
* Patients who received rituximab or amifostine within 30 days prior to first telmisartan dose on this study
* Patients on ramapril
* Patients on digoxin who do not consent to monthly digoxin blood level testing

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Tolerability of oral telmisartan | 12 months
  Ability of the participant to tolerate telmisartan alone or with standard of care agents as defined by maintaining a systolic blood pressure >110mmHG and are without greater than grade 2 toxicities

SECONDARY OUTCOMES:
Increase in tumor DNA damage | 24 months
  Determine if telmisartan increases tumor DNA damage or alters immunity in ways consistent with anti-tumor activity when given alone or with selected standard of care treatments in selected patients with prostate cancer as determined by counting gamma-H2AX foci in tissue sections and peripheral blood mononuclear cells

OTHER OUTCOMES:
Reduction of blood prostate specific antigen | 24 months
  This exploratory objective is to determine whether telmisartan when given alone or combined with selected standard of care therapies can reduce blood prostate specific antigen or slow its rise in selected patients with prostate cancer as determined by Roche Cobas immunoassay in ng/mL blood

CONTACTS AND LOCATIONS:
Overall Officials: Rodwell Mabaera, MD, Principal Investigator — Dartmouth Health
Locations (1):
- Dartmouth Health, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] SEER*Explorer: An interactive website for SEER cancer statistics [Internet]. Surveillance Research Program, National Cancer Institute; 2023 Apr 19. Available from: https://seer.cancer.gov/statistics-network/explorer/. Data source(s): SEER Incidence Data, November 2022 Submission (1975-2020), SEER 22 registries. updated: 2023 Jun 8. Accessed Oct 5, 2023
- [Background] Smith MR, Saad F, Rathkopf DE, Mulders PFA, de Bono JS, Small EJ, Shore ND, Fizazi K, Kheoh T, Li J, De Porre P, Todd MB, Yu MK, Ryan CJ. Clinical Outcomes from Androgen Signaling-directed Therapy after Treatment with Abiraterone Acetate and Prednisone in Patients with Metastatic Castration-resistant Prostate Cancer: Post Hoc Analysis of COU-AA-302. Eur Urol. 2017 Jul;72(1):10-13. doi: 10.1016/j.eururo.2017.03.007. Epub 2017 Mar 15. PMID 28314611
- [Background] Chen K, O'Brien J, McVey A, Jenjitranant P, Kelly BD, Kasivisvanathan V, Lawrentschuk N, Murphy DG, Azad AA. Combination treatment in metastatic prostate cancer: is the bar too high or have we fallen short? Nat Rev Urol. 2023 Feb;20(2):116-123. doi: 10.1038/s41585-022-00669-z. Epub 2022 Dec 12. PMID 36509970
- [Background] Sayegh N, Swami U, Agarwal N. Recent Advances in the Management of Metastatic Prostate Cancer. JCO Oncol Pract. 2022 Jan;18(1):45-55. doi: 10.1200/OP.21.00206. Epub 2021 Sep 2. PMID 34473525
- [Background] Asim M, Tarish F, Zecchini HI, Sanjiv K, Gelali E, Massie CE, Baridi A, Warren AY, Zhao W, Ogris C, McDuffus LA, Mascalchi P, Shaw G, Dev H, Wadhwa K, Wijnhoven P, Forment JV, Lyons SR, Lynch AG, O'Neill C, Zecchini VR, Rennie PS, Baniahmad A, Tavare S, Mills IG, Galanty Y, Crosetto N, Schultz N, Neal D, Helleday T. Synthetic lethality between androgen receptor signalling and the PARP pathway in prostate cancer. Nat Commun. 2017 Aug 29;8(1):374. doi: 10.1038/s41467-017-00393-y. PMID 28851861
- [Background] Saad F, Clarke NW, Oya M, Shore N, Procopio G, Guedes JD, Arslan C, Mehra N, Parnis F, Brown E, Schlurmann F, Joung JY, Sugimoto M, Sartor O, Liu YZ, Poehlein C, Barker L, Del Rosario PM, Armstrong AJ. Olaparib plus abiraterone versus placebo plus abiraterone in metastatic castration-resistant prostate cancer (PROpel): final prespecified overall survival results of a randomised, double-blind, phase 3 trial. Lancet Oncol. 2023 Oct;24(10):1094-1108. doi: 10.1016/S1470-2045(23)00382-0. Epub 2023 Sep 12. PMID 37714168
- [Background] Murray C, Bai H, Ontiveros CO, et al. Pharmacologic tumor PDL1 depletion as a novel approach to overcome treatment resistance. The Journal of Immunology. 2023;210(1_Supplement):230.08-230.08. doi:10.4049/jimmunol.210.Supp.230.08
- [Background] Uemura H, Miyoshi Y, Ishiguro H, Nakaigawa N, Noguchi K, Kubota Y. Effectiveness of angionten II receptor blocker (ARB), candesartan, in the treatment of hormone refractory prostate cancer (HRPC). presented at: 2004 ASCO Annual Meeting; 2004
- [Background] Wang C, Wang WB. Telmisartan Induces Osteosarcoma Cells Growth Inhibition and Apoptosis Via Suppressing mTOR Pathway. Open Life Sci. 2018 Jul 5;13:242-249. doi: 10.1515/biol-2018-0029. eCollection 2018 Jan. PMID 33817089
- [Background] Scher HI, Morris MJ, Stadler WM, Higano C, Basch E, Fizazi K, Antonarakis ES, Beer TM, Carducci MA, Chi KN, Corn PG, de Bono JS, Dreicer R, George DJ, Heath EI, Hussain M, Kelly WK, Liu G, Logothetis C, Nanus D, Stein MN, Rathkopf DE, Slovin SF, Ryan CJ, Sartor O, Small EJ, Smith MR, Sternberg CN, Taplin ME, Wilding G, Nelson PS, Schwartz LH, Halabi S, Kantoff PW, Armstrong AJ; Prostate Cancer Clinical Trials Working Group 3. Trial Design and Objectives for Castration-Resistant Prostate Cancer: Updated Recommendations From the Prostate Cancer Clinical Trials Working Group 3. J Clin Oncol. 2016 Apr 20;34(12):1402-18. doi: 10.1200/JCO.2015.64.2702. Epub 2016 Feb 22. PMID 26903579
- [Background] Jensterle M, Janez A, Vrtovec B, Meden-Vrtovec H, Pfeifer M, Prezelj J, Kocjan T. Decreased androgen levels and improved menstrual pattern after angiotensin II receptor antagonist telmisartan treatment in four hypertensive patients with polycystic ovary syndrome: case series. Croat Med J. 2007 Dec;48(6):864-70. doi: 10.3325/cmj.2007.6.864. PMID 18074422
- [Background] McAlister FA; Renin Angiotension System Modulator Meta-Analysis Investigators. Angiotensin-converting enzyme inhibitors or angiotensin receptor blockers are beneficial in normotensive atherosclerotic patients: a collaborative meta-analysis of randomized trials. Eur Heart J. 2012 Feb;33(4):505-14. doi: 10.1093/eurheartj/ehr400. Epub 2011 Oct 31. PMID 22041554
- [Background] Galle J. Reduction of proteinuria with angiotensin receptor blockers. Nat Clin Pract Cardiovasc Med. 2008 Jul;5 Suppl 1:S36-43. doi: 10.1038/ncpcardio0806. PMID 18580865
- [Background] Qaisar R, Kamli H, Karim A, Muhammad T, Ahmad F, Shaikh A. Angiotensin Receptor Blockers Restore Skeletal Muscle in Patients with Chronic Obstructive Pulmonary Disease. Arch Med Res. 2023 Nov;54(7):102890. doi: 10.1016/j.arcmed.2023.102890. Epub 2023 Sep 21. PMID 37741098
- [Background] Fang T, Zhang J, Zuo T, Wu G, Xu Y, Yang Y, Yang J, Shen Q. Chemo-Photothermal Combination Cancer Therapy with ROS Scavenging, Extracellular Matrix Depletion, and Tumor Immune Activation by Telmisartan and Diselenide-Paclitaxel Prodrug Loaded Nanoparticles. ACS Appl Mater Interfaces. 2020 Jul 15;12(28):31292-31308. doi: 10.1021/acsami.0c10416. Epub 2020 Jul 1. PMID 32551473
- [Background] Zhu Y, Yu F, Tan Y, Hong Y, Meng T, Liu Y, Dai S, Qiu G, Yuan H, Hu F. Reversing activity of cancer associated fibroblast for staged glycolipid micelles against internal breast tumor cells. Theranostics. 2019 Sep 19;9(23):6764-6779. doi: 10.7150/thno.36334. eCollection 2019. PMID 31660067
- [Background] Kobara H, Fujihara S, Iwama H, Matsui T, Fujimori A, Chiyo T, Tingting S, Kobayashi N, Nishiyama N, Yachida T, Tadokoro T, Oura K, Tani J, Fujita K, Nomura T, Yoneyama H, Morishita A, Okano K, Suzuki Y, Mori H, Masaki T. Antihypertensive drug telmisartan inhibits cell proliferation of gastrointestinal stromal tumor cells in vitro. Mol Med Rep. 2020 Aug;22(2):1063-1071. doi: 10.3892/mmr.2020.11144. Epub 2020 May 14. PMID 32626983
- [Background] Fujita N, Fujita K, Iwama H, Kobara H, Fujihara S, Chiyo T, Namima D, Yamana H, Kono T, Takuma K, Hirata M, Kobayashi K, Kato K, Kamada H, Morishita A, Tsutsui K, Himoto T, Okano K, Suzuki Y, Masaki T. Antihypertensive drug telmisartan suppresses the proliferation of gastric cancer cells in vitro and in vivo. Oncol Rep. 2020 Jul;44(1):339-348. doi: 10.3892/or.2020.7607. Epub 2020 May 7. PMID 32627043
- [Background] Uemura H, Ishiguro H, Nakaigawa N, Nagashima Y, Miyoshi Y, Fujinami K, Sakaguchi A, Kubota Y. Angiotensin II receptor blocker shows antiproliferative activity in prostate cancer cells: a possibility of tyrosine kinase inhibitor of growth factor. Mol Cancer Ther. 2003 Nov;2(11):1139-47. PMID 14617787
- [Background] Wu TT, Niu HS, Chen LJ, Cheng JT, Tong YC. Increase of human prostate cancer cell (DU145) apoptosis by telmisartan through PPAR-delta pathway. Eur J Pharmacol. 2016 Mar 15;775:35-42. doi: 10.1016/j.ejphar.2016.02.017. Epub 2016 Feb 4. PMID 26852954
- [Background] Takahashi S, Uemura H, Seeni A, Tang M, Komiya M, Long N, Ishiguro H, Kubota Y, Shirai T. Therapeutic targeting of angiotensin II receptor type 1 to regulate androgen receptor in prostate cancer. Prostate. 2012 Oct 1;72(14):1559-72. doi: 10.1002/pros.22505. Epub 2012 Mar 16. PMID 22430461
- [Background] Mariniello M, Petruzzelli R, Wanderlingh LG, La Montagna R, Carissimo A, Pane F, Amoresano A, Ilyechova EY, Galagudza MM, Catalano F, Crispino R, Puchkova LV, Medina DL, Polishchuk RS. Synthetic Lethality Screening Identifies FDA-Approved Drugs that Overcome ATP7B-Mediated Tolerance of Tumor Cells to Cisplatin. Cancers (Basel). 2020 Mar 6;12(3):608. doi: 10.3390/cancers12030608. PMID 32155756
- [Background] Green R, Howell M, Khalil R, Nair R, Yan J, Foran E, Katiri S, Banerjee J, Singh M, Bharadwaj S, Mohapatra SS, Mohapatra S. Actinomycin D and Telmisartan Combination Targets Lung Cancer Stem Cells Through the Wnt/Beta Catenin Pathway. Sci Rep. 2019 Dec 3;9(1):18177. doi: 10.1038/s41598-019-54266-z. PMID 31796785
- [Background] Rasheduzzaman M, Moon JH, Lee JH, Nazim UM, Park SY. Telmisartan generates ROS-dependent upregulation of death receptor 5 to sensitize TRAIL in lung cancer via inhibition of autophagy flux. Int J Biochem Cell Biol. 2018 Sep;102:20-30. doi: 10.1016/j.biocel.2018.06.006. Epub 2018 Jun 19. PMID 29929000
- [Background] Grahovac J, Srdic-Rajic T, Francisco Santibanez J, Pavlovic M, Cavic M, Radulovic S. Telmisartan induces melanoma cell apoptosis and synergizes with vemurafenib in vitro by altering cell bioenergetics. Cancer Biol Med. 2019 May;16(2):247-263. doi: 10.20892/j.issn.2095-3941.2018.0375. PMID 31516746
- [Background] Samukawa E, Fujihara S, Oura K, Iwama H, Yamana Y, Tadokoro T, Chiyo T, Kobayashi K, Morishita A, Nakahara M, Kobara H, Mori H, Okano K, Suzuki Y, Himoto T, Masaki T. Angiotensin receptor blocker telmisartan inhibits cell proliferation and tumor growth of cholangiocarcinoma through cell cycle arrest. Int J Oncol. 2017 Dec;51(6):1674-1684. doi: 10.3892/ijo.2017.4177. Epub 2017 Oct 23. PMID 29075786
- [Background] Oura K, Tadokoro T, Fujihara S, Morishita A, Chiyo T, Samukawa E, Yamana Y, Fujita K, Sakamoto T, Nomura T, Yoneyama H, Kobara H, Mori H, Iwama H, Okano K, Suzuki Y, Masaki T. Telmisartan inhibits hepatocellular carcinoma cell proliferation in vitro by inducing cell cycle arrest. Oncol Rep. 2017 Nov;38(5):2825-2835. doi: 10.3892/or.2017.5977. Epub 2017 Sep 20. PMID 29048654
- [Background] Fujihara S, Morishita A, Ogawa K, Tadokoro T, Chiyo T, Kato K, Kobara H, Mori H, Iwama H, Masaki T. The angiotensin II type 1 receptor antagonist telmisartan inhibits cell proliferation and tumor growth of esophageal adenocarcinoma via the AMPKalpha/mTOR pathway in vitro and in vivo. Oncotarget. 2017 Jan 31;8(5):8536-8549. doi: 10.18632/oncotarget.14345. PMID 28052030
- [Background] Pu Z, Zhu M, Kong F. Telmisartan prevents proliferation and promotes apoptosis of human ovarian cancer cells through upregulating PPARgamma and downregulating MMP-9 expression. Mol Med Rep. 2016 Jan;13(1):555-9. doi: 10.3892/mmr.2015.4512. Epub 2015 Nov 6. PMID 26548340
- [Background] de Araujo Junior RF, Leitao Oliveira AL, de Melo Silveira RF, de Oliveira Rocha HA, de Franca Cavalcanti P, de Araujo AA. Telmisartan induces apoptosis and regulates Bcl-2 in human renal cancer cells. Exp Biol Med (Maywood). 2015 Jan;240(1):34-44. doi: 10.1177/1535370214546267. Epub 2014 Aug 14. PMID 25125501
- [Background] Ozeki K, Tanida S, Morimoto C, Inoue Y, Mizoshita T, Tsukamoto H, Shimura T, Kataoka H, Kamiya T, Nishiwaki E, Ishiguro H, Higashiyama S, Joh T. Telmisartan inhibits cell proliferation by blocking nuclear translocation of ProHB-EGF C-terminal fragment in colon cancer cells. PLoS One. 2013;8(2):e56770. doi: 10.1371/journal.pone.0056770. Epub 2013 Feb 22. PMID 23451083
- [Background] Koyama N, Nishida Y, Ishii T, Yoshida T, Furukawa Y, Narahara H. Telmisartan induces growth inhibition, DNA double-strand breaks and apoptosis in human endometrial cancer cells. PLoS One. 2014 Mar 25;9(3):e93050. doi: 10.1371/journal.pone.0093050. eCollection 2014. PMID 24667764
- [Background] Kornepati AVR, Boyd JT, Murray CE, Saifetiarova J, de la Pena Avalos B, Rogers CM, Bai H, Padron AS, Liao Y, Ontiveros C, Svatek RS, Hromas R, Li R, Hu Y, Conejo-Garcia JR, Vadlamudi RK, Zhao W, Dray E, Sung P, Curiel TJ. Tumor Intrinsic PD-L1 Promotes DNA Repair in Distinct Cancers and Suppresses PARP Inhibitor-Induced Synthetic Lethality. Cancer Res. 2022 Jun 6;82(11):2156-2170. doi: 10.1158/0008-5472.CAN-21-2076. PMID 35247877
- [Background] Nair AB, Jacob S. A simple practice guide for dose conversion between animals and human. J Basic Clin Pharm. 2016 Mar;7(2):27-31. doi: 10.4103/0976-0105.177703. PMID 27057123
- [Background] Daniel B, Nagy G, Czimmerer Z, Horvath A, Hammers DW, Cuaranta-Monroy I, Poliska S, Tzerpos P, Kolostyak Z, Hays TT, Patsalos A, Houtman R, Sauer S, Francois-Deleuze J, Rastinejad F, Balint BL, Sweeney HL, Nagy L. The Nuclear Receptor PPARgamma Controls Progressive Macrophage Polarization as a Ligand-Insensitive Epigenomic Ratchet of Transcriptional Memory. Immunity. 2018 Oct 16;49(4):615-626.e6. doi: 10.1016/j.immuni.2018.09.005. PMID 30332629
- [Background] Kornepati AVR, Rogers CM, Sung P, Curiel TJ. The complementarity of DDR, nucleic acids and anti-tumour immunity. Nature. 2023 Jul;619(7970):475-486. doi: 10.1038/s41586-023-06069-6. Epub 2023 Jul 19. PMID 37468584
- [Background] Washida K, Ihara M, Nishio K, Fujita Y, Maki T, Yamada M, Takahashi J, Wu X, Kihara T, Ito H, Tomimoto H, Takahashi R. Nonhypotensive dose of telmisartan attenuates cognitive impairment partially due to peroxisome proliferator-activated receptor-gamma activation in mice with chronic cerebral hypoperfusion. Stroke. 2010 Aug;41(8):1798-806. doi: 10.1161/STROKEAHA.110.583948. Epub 2010 Jul 1. PMID 20595663
- [Background] Torika N, Asraf K, Danon A, Apte RN, Fleisher-Berkovich S. Telmisartan Modulates Glial Activation: In Vitro and In Vivo Studies. PLoS One. 2016 May 17;11(5):e0155823. doi: 10.1371/journal.pone.0155823. eCollection 2016. PMID 27187688
- [Background] Hartley A, Ahmad I. The role of PPARgamma in prostate cancer development and progression. Br J Cancer. 2023 Apr;128(6):940-945. doi: 10.1038/s41416-022-02096-8. Epub 2022 Dec 12. PMID 36510001
- [Background] Khorsand M, Khajeh S, Eslami M, Nezafat N, Ghasemi Y, Razban V, Mostafavi-Pour Z. Telmisartan anti-cancer activities mechanism through targeting N-cadherin by mimicking ADH-1 function. J Cell Mol Med. 2022 Apr;26(8):2392-2403. doi: 10.1111/jcmm.17259. Epub 2022 Feb 27. PMID 35224849
- [Background] Cernes R, Mashavi M, Zimlichman R. Differential clinical profile of candesartan compared to other angiotensin receptor blockers. Vasc Health Risk Manag. 2011;7:749-59. doi: 10.2147/VHRM.S22591. Epub 2011 Dec 12. PMID 22241949
- [Background] Uemura H, Hasumi H, Kawahara T, Sugiura S, Miyoshi Y, Nakaigawa N, Teranishi J, Noguchi K, Ishiguro H, Kubota Y. Pilot study of angiotensin II receptor blocker in advanced hormone-refractory prostate cancer. Int J Clin Oncol. 2005 Dec;10(6):405-10. doi: 10.1007/s10147-005-0520-y. PMID 16369744
- [Background] Funao K, Matsuyama M, Kawahito Y, Sano H, Chargui J, Touraine JL, Nakatani T, Yoshimura R. Telmisartan is a potent target for prevention and treatment in human prostate cancer. Oncol Rep. 2008 Aug;20(2):295-300. PMID 18636189
- [Background] Uemura H, Kubota Y. [Application of angiotensin II receptor blocker in prostate cancer]. Nihon Rinsho. 2009 Apr;67(4):807-11. Japanese. PMID 19348246
- [Background] Tascilar K, Azoulay L, Dell'Aniello S, Bartels DB, Suissa S. The Use of Telmisartan and the Incidence of Cancer. Am J Hypertens. 2016 Dec 1;29(12):1358-1365. doi: 10.1093/ajh/hpw095. PMID 27557862
- [Background] Wilk M, Wasko-Grabowska A, Skoneczna I, Szmit S. Angiotensin System Inhibitors May Improve Outcomes of Patients With Castration-Resistant Prostate Cancer During Abiraterone Acetate Treatment-A Cardio-Oncology Study. Front Oncol. 2021 Apr 1;11:664741. doi: 10.3389/fonc.2021.664741. eCollection 2021. PMID 33869068
- [Background] Rudolph J, Jung K, Luger K. Inhibitors of PARP: Number crunching and structure gazing. Proc Natl Acad Sci U S A. 2022 Mar 15;119(11):e2121979119. doi: 10.1073/pnas.2121979119. Epub 2022 Mar 8. PMID 35259019
- [Background] LaFargue CJ, Dal Molin GZ, Sood AK, Coleman RL. Exploring and comparing adverse events between PARP inhibitors. Lancet Oncol. 2019 Jan;20(1):e15-e28. doi: 10.1016/S1470-2045(18)30786-1. PMID 30614472